CLINICAL TRIAL: NCT06235047
Title: Liposomal Doxorubicin-containing Front-line Treatment in Elderly Patients With Classic Hodgkin Lymphoma: a Multicenter Phase II Study
Brief Title: Liposomal Doxorubicin-containing Front-line Treatment in Elderly Patients With HL (HL-MVD)
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Professor, Federico II University
Other Study IDs: FED-HL-MVD
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Classic Hodgkin Lymphoma
Keywords: cHL; >60y; liposomal doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on the use of a polychemotherapy scheme based on liposomal doxorubicin, vinblastine and dacarbazine (MVD) as first line in the therapy of elderly patients affected by classic Hodgkin lymphoma

DETAILED DESCRIPTION:
Classic Hodgkin lymphoma (c-HL) is a neoplasm that originates from B lymphocytes and represents 10% of all lymphomas. The most affected age group is between 20 and 30 years of age, with a second peak in the epidemiological distribution involving patients over 60 years of age.

Elderly patients often present with already advanced disease stages and B symptoms. On the other hand, these patients often have multiple comorbidities and reduced fitness and this can limit the therapeutic possibilities with curative intent in terms of doses and adherence to the timing foreseen by the therapeutic protocol.

The optimal therapy for this category of patients is not yet well defined. In fact, the prognosis of these patients is typically poor.

The ABVD regimen (doxorubicin, i.e. Adriamycin, Bleomycin, Vinblastine, Dacarbazine) is a therapeutic option for elderly/unfit patients but is associated with considerable toxicity and mortality. In particular, mortality rates due to lung damage from Bleomycin are between 4-24% and mortality rates due to cardiac damage are reported in elderly patients suffering from c-HL and treated with regimens based on anthracyclines (of which doxorubicin belongs part) which fluctuate between 6 and 15%.

Non-pegylated liposomal anthracycline (NPLD) was initially used in patients with breast cancer and this particular formulation spares tissues characterized by tight capillary junctions (such as cardiac muscle tissue) from the direct cytotoxic effect of doxorubicin.

Regimens based on NPLD associated with bleomycin, vinblastine and dacarbazine have been studied for the first-line treatment of cardiac patients with c-HL and NPLD has been shown to accumulate in macrophages associated with tumor tissue, as well as in the spleen, liver, lung and bones that act as long-release reservoirs with a likely prolonged therapeutic effect.

The aim of the present project is to investigate the front-line use of the MVD polychemotherapeutic regimen (NPLD, Bleomycin and Dacarbazine) for elderly patients suffering from c-HL in terms of Overall Survival, Progression-Free Survival, FDG-PET/CT negativity rate at the end of therapy, toxicity and feasibility.

This was a retrospective, single-center study conducted in the Hematology Unit of the Federico II University of Naples (Italy), in which patients aged ≥60 years with previously untreated, biopsy-proven c-HL were identified in the database of the Hematology Unit of the Federico II University from 1 January 2013 to 1 January 2023. All necessary approvals were obtained from our ethics committee. The study was undertaken in accordance with the Declaration of Helsinki. All patients provided written informed consent for data analysis.

The primary objective of the study was to evaluate whether the front-line therapy without bleomycin by using NPLD-containing regimen, i.e., Myocet TM with its pharmacokinetic and pharmacodynamic advantages in terms of efficacy and safety, could improve OS in older adults with c-HL with extensive disease. Other objectives were PFS, EoT overall response rate by using FDG-PET scans interpreted with the Deauville scale (DS) 5-point scoring system (according to the Lugano Classification) , hematologic and extra-hematologic toxicity (according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0), and feasibility (arbitrarily defined as ≤5 patients receiving <85% of the planned dose). Noteworthy, the cardiologic toxicity profile was established by using the echocardiography assessment of global systolic longitudinal myocardial strain (GLS), as well as left ventricular ejection fraction (LVEF) (according to the guidelines of the Task Force for Cancer Treatments and Cardiovascular Toxicity of the European Society of Cardiology [ESC]).

The schedule of study treatment is shown in detail in Table 1. The dosage of Myocet TM in the MVD scheme was well within the ceiling dose of 785 mg/m 2 (the median lifetime dose reported for NPLD at the onset of cardiotoxicity). Patients were scheduled to receive six cycles of therapy with MVD which consisted of 1-day outpatient i.v. infusions of Myocet TM at a dose of 25 mg/m 2 , plus vinblastine 6 mg/m 2 , and dacarbazine 375 mg/m 2 on days 1 and 14 of each course every 28 days, for twelve administrations. Planned cumulative dose-intensity of NPLD was 300 mg/m 2.

For those cases with initial large nodal mass (defined as systemic adenopathy with the largest diameter >5 cm), consolidation radiotherapy (c-RT) at 30 Gy was given (after EoT PET assessments), following the scheduled 6 MVD cycles, on residual bulky area, that is, containing post-chemotherapy FDG-PET negative nodes of size ≥2.0 cm at CT scans as already reported.

FDG-PET examinations were conducted at staging, EoT and thereafter every 3-6 months. FDG-PET results were reported according to the DS score using visual assessment followed by quantitative verification as already described. Negative FDG-PET scans were defined as DS ≤3 score, and positive FDG-PET scans were defined as DS 4 and 5 scores (Supplemental data, FDG- PET assessments). All patients were scheduled to undergo a full cardiologic examination, 2D echocardiography, and speckle tracking echocardiography (STE) at baseline, interim, EoT and within six months from the end of all antineoplastic treatments.

Clinical cardiologist experts in echocardiography analyzed each study for standard echocardiography and strain measurements.

Physical examination and bone marrow biopsy were also performed at baseline, and then at physician's discretion. Routine blood laboratory test monitoring was performed before every cycle of chemotherapy, for each patient.

OS was defined as the time from the date of HL diagnosis to the date of last follow-up or death for any cause. PFS was defined as the time from day 1 of MVD ﬁrst dose to disease progression/relapse (event), death from any cause (event) or last follow-up visit (censoring). All efficacy and safety evaluations were performed in patients who received at least one course of MVD. Patients' characteristics, response rate, toxicity and safety data were reported descriptively as number and percentage, or as median and range. Survival curves were estimated by the Kaplan-Meier method. Cox regression analysis was used to estimate the hazard ratio (HR) and the 95% confidence interval (CI) for the treatment effect on OS and PFS. The evaluated factors included age stratification (years: 60-69 vs. 70-79 vs. ≥80), B symptoms, large nodal mass, nodal and/or extra-nodal sites involved, stage IV, and international prognostic score (IPS) risk group at baseline. Differences between groups were tested by the log-rank test, and student-T test. The P value for statistical significance was set at 0.05 for all evaluations. Statistical analysis was performed using R software (version 4.1).

ELIGIBILITY:
Inclusion Criteria:

* previously untreated, biopsy-proven c-HL
* Ann Arbor stage III or IV
* ECOG PS 0-3
* LVEF≥50% at echocardiographic assessment
* human immunodeficiency virus negativity.
* any GLS value

Exclusion Criteria:

* Ann Arbor stage I or II,
* concomitant major illnesses
* creatinine clearance <30 ml/min
* serum transaminases more than three times the normal value
* total bilirubin >3.4 mg/dl
* absolute neutrophil count <500/mm 3
* hemoglobin level <9 g/dL
* platelet count <75 000/mm 3
* Myocardial infarction represented an exclusion only if diagnosed within 3 months prior to MVD start.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: over60 year old c-HL patients, previously untreated with Ann Arbor stage III or IV. ECOG PS 0-3, GLS ≥-20% at echocardiographic assessment and human immunodeficiency virus negativity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | from 1 January 2013 to 1 January 2023
  The primary endpoint was the activity of the liposomal doxorubicin-based front-line strategy in terms of OS.

SECONDARY OUTCOMES:
Progression-free survival | from 1 January 2013 to 1 January 2023
  Progression free survival
End of Treatment response rate | from 1 January 2013 to 1 January 2023
  end-of-treatment (EoT) 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography (FDG-PET)-negativity
Adverse events | from 1 January 2013 to 1 January 2023
  hematological and cardiac grade >3 adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy